CLINICAL TRIAL: NCT06375044
Title: A Phase I First-in-human, Open-label Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0500, A Humanized GPRC5D-BCMA-CD3 Tri-specific Antibody, in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of SIM0500 Alone in Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0500-101
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SIM0500 (Experimental)
  Interventions: Drug: SIM0500

INTERVENTIONS:
Drug: SIM0500 — Participants will receive SIM0500 in a 28-day cycle until disease progression, intolerable toxicity, or until the participant voluntarily withdraws from trial intervention, or end of study, whichever comes first.

SUMMARY:
This is an open-label, multicenter phase 1 clinical trial to evaluate the safety and tolerability, efficacy, and pharmacokinetics of SIM0500 in adult participants with Relapsed or Refractory Multiple Myeloma(RRMM). The trial is consisted of two parts, Part 1 (dose escalation) and Part 2 (dose optimization). In both parts, SIM0500 will be administered until disease progression, intolerable toxicity, withdraw of consent or end of trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent form.
2. ≥18 years of age.
3. Have documented diagnosis of relapsed or refractory multiple myeloma according to Criteria for Response to Multiple Myeloma Treatment(IMWG)diagnostic criteria who have failed all established standard of care.
4. Life expectancy ≥12 weeks.
5. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
6. Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

1. Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy.
2. Active hepatitis B (HBsAg positive and HBV DNA ≥ 1×104 copies/mL or ≥ 2,000 international unit [IU]/mL) or hepatitis C (HCV antibody positive and HCV RNA ≥ ULN) infection; participant with HBsAg positive or detective HBV-DNA at screening should receive antiviral treatment as per local practice during the trial.
3. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
4. Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
5. Active known or suspected autoimmune disease. Participants with vitiligo, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger, type 1 diabetes mellitus (blood glucose can be controlled by insulin therapy) can be included.
6. Current or previous other malignancy within 3 years of study entry, except basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast.
7. Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
8. Participants with known active infection within 14 days prior to the first SIM0500.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Dana Farber Cancer institution, Boston, Massachusetts
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai，The Tisch Cancer Institute, New York, New York
- China (5):
  - Beijing Chaoyang Hospital Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hanzhou, Zhejiang